CLINICAL TRIAL: NCT00571662
Title: Allogeneic Peripheral Blood Stem Cell Transplantation With Minimally Myelosuppressive Regimen of Pentostatin and Low-dose Total-body Irradiation
Brief Title: Safety and Efficacy of Pentostatin and Low Dose TBI With Allogenic Peripheral Blood Stem Cell Transplant
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: Astex Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0389-00-FB
Record Dates: First submitted 2007-12-11; First posted 2007-12-12 (Estimated); Results first posted 2010-11-17 (Estimated); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Acute Myelogenous Leukemia; Acute Lymphocytic Leukemia; Chronic Myelogenous Leukemia; Chronic Lymphocytic Leukemia; Myelodysplastic Syndromes; Multiple Myeloma; Non-Hodgkins Lymphoma; Hodgkins Disease; Peripheral T-cell Lymphoma
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Lymphocytic, Chronic, B-Cell; Myelodysplastic Syndromes; Multiple Myeloma; Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma, T-Cell, Peripheral | interventions — Pentostatin; Whole-Body Irradiation; Cyclosporine; Mycophenolic Acid; Granulocyte Colony-Stimulating Factor; sargramostim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cohort I (Experimental): Pentostatin to be administered intravenously on days - 10, -9, and -8 at a dose of 4mg/m2/day
  Interventions: Drug: Pentostatin; Radiation: Total-body irradiation (TBI); Drug: Cyclosporine A (CsA); Drug: Mycophenolate Mofetil (MMF); Drug: G-CSF

INTERVENTIONS:
Drug: Pentostatin — 4 mg/m^2 intravenous(IV)once a day(QD)x3days (days -10, -9, -8)
  Other Names: Nipent
Radiation: Total-body irradiation (TBI) — TBI will consist of 2.0 GY at 8-12cGy/min via 6MV photons delivered AP/PA fields, without lung blocks or via lateral fields with lucite compensator along the head and neck region. TLD (thermal luminescent dosimetry) will be used to verify dose uniformity. TBI will be given on day -1.
Drug: Cyclosporine A (CsA) — CsA will be given at 2.0 mg/kg intravenous (IV) Q 12hrs on days -1,0,and+1 (total 6 doses) then converted to oral at 2 mg/kg by mouth (PO) twice a day (BID) until day+80, then tapered 10% per week over approximately 3 months if no GVHD for related donor transplants. For unrelated CsA will be given at same dose and schedule until day+100 then tapered by 10% per week if no GVHD
  Other Names: Neoral
Drug: Mycophenolate Mofetil (MMF) — MMF 15 mg/kg by mouth twice a day (PO BID) will be given from day 0-27 then stopped without tapering for related donor transplants. For unrelated donor transplants MMF will be given at same dose until day+40 then tapered over 2months. in absence of GVHD. Doses will be rounded to nearest 250 mg.
Drug: G-CSF — 10 mcg/kg/day subcutaneously for at least 4 consecutive days.
  Other Names: Leukine

SUMMARY:
This is a continuation of a pilot study which is now regarded as a phase II trial with a plan to enroll an additional 40 patients (20 related and 20 unrelated donor transplants) with hematological malignancy assessing the safety and efficacy of a minimally myelosuppressive regimen with pentostatin and low-dose total body irradiation (TBI) followed by allogeneic peripheral blood stem cell transplantation (alloPSCT).

DETAILED DESCRIPTION:
This is a pilot study which began with a plan to enroll 50 patients (20 related and 30 unrelated donor transplants) with hematological malignancy assessing the safety and efficacy of a minimally myelosuppressive regimen with Pentostatin and low-dose total body irradiation (TBI) followed by allogeneic peripheral blood stem cell transplantation (alloPSCT). Patients with persistent or progressive malignancy after transplantation will be treated with GM-CSF (cytokine therapy) to assess its toxicity and potential therapeutic efficacy. Patients with persistent or progressive disease who fail or do not qualify for the cytokine therapy portion of the study will become candidates for donor leukocyte infusions.

The purpose of this protocol remains a pilot study which is now regarded as a phase II trial with a plan to enroll 40 ADDITIONAL patients (20 related and 20 unrelated donor transplants) with hematological malignancy assessing the safety and efficacy of a modified version of the original preparative regimen of Pentostatin and low-dose total body irradiation (TBI) followed by allogeneic peripheral blood stem cell transplantation (alloPSCT). Patients who fail will become candidates for donor-leukocyte infusion (DLI).

Primary Objectives

1. To determine the safety of treating hematological malignancies by establishing donor hematopoietic chimerism using pentostatin and low-dose total body irradiation followed by allogeneic peripheral blood stem cell transplantation.
2. To determine the immunomodulatory effects of pentostatin as part of the conditioning regimen for allogeneic peripheral blood stem cell transplantation.

Secondary Objectives

1. To determine the incidence of infections after using a minimally myelosuppressive conditioning regimen.
2. To determine the kinetics of hematological and immunological reconstitution after allotransplantation with a minimally myelosuppressive conditioning regimen.
3. To determine the incidence of chronic GVHD after using allogeneic peripheral blood stem cell transplantation with a minimally myelosuppressive preparative regimen.
4. To evaluate the role of the preparative regimen and donor source (related versus unrelated) on inflammatory cytokine profiles.
5. To evaluate blood and where possible, biopsy specimens for a recently identified nuclear protein (molecular weight 44/46) in mononuclear cells obtained from study subjects.

Interventions, evaluation, and follow up will include:

Pentostatin 4 mg/m^2/d intravenously once a day x 3 days will be administered with 1000 cc NS hydration before and after pentostatin ten days prior to stem cell infusion (days -10, -9, and -8). Total-body irradiation (TBI): TBI 2.0 Gy will be given on day -1. Antiemetics will be given as needed. Patients will receive one liter normal saline over 2 hours pre TBI. A bone marrow biopsy and aspiration with cytogenetics and flow cytometry will be performed on Day +28, Day +70 and 6, 12, 18 and 24 months following the transplant to monitor hematologic recovery. DNA fingerprinting will also be conducted at the same time at 3, 4, 5, 6, 12, 18, and 24 months to determine chimerism.

ELIGIBILITY:
Inclusion Criteria:

Age 19-75 years

1. Patients who relapse after autologous stem cell transplantation.
2. Patients who are candidates for an autologous or conventional allogeneic stem cell transplantation from a disease standpoint but who do not qualify functionally (from the point of view of organ function, or performance status) for a myeloablative protocol.
3. Any patient, where in the opinion of the primary treating oncologist, nonmyleoablative therapy would be the treatment option in the best patients interest providing the patient fits all other eligibility criteria for this protocol.

Identification of a matched related or unrelated stem cell donor

Diseases:

Acute myelogenous leukemia first complete remission with high-risk cytogenetics>second complete remission minimal residual disease (<10% blasts*). Acute lymphocytic leukemia first complete remission with high-risk cytogenetics >second complete remission minimal residual disease (<10% blasts*). Chronic myelogenous leukemia first chronic phase, accelerated phase (<10% blasts*)blast phase with minimal residual disease (<10% blasts*)second chronic phase. Chronic lymphocytic leukemia recurrence after the front line regimen (related donor transplant), chemorefractory disease (unrelated donor transplant),T-CLL in partial remission or any minimal residual disease. Myelodysplastic syndromes refractory anemia with or without ringed sideroblasts,RAEB, RAEB-T, and CMML (< than 10% blasts*). *both in peripheral blood and bone marrow

Multiple myeloma - after receiving at least one regimen of prior chemotherapy

Non-Hodgkin's Lymphomas:

Small Lympho(plasma)cytic Lymphoma (B-SLL, B-LPL): recurrence after a front line regimen (related donor transplant), or chemorefractory disease (related or unrelated donor transplant). Follicular Low-Grade Lymphoma, Marginal Zone Lymphomas (splenic, nodal, or extranodal/MALT type): chemorefractory disease or > 2 prior regimens. Mantle Cell Lymphoma: first complete or partial remission, refractory disease, or failed prior ASCT. Diffuse Large B-cell Lymphoma, Follicular Large cell Lymphoma, Peripheral T-cell Lymphoma, Anaplastic Large Cell Lymphoma: refractory disease, or failed prior ASCT. Burkitt or Acute Lymphoblastic Lymphomas: high-risk disease in remission, chemosensitive persistent or recurrent disease. Cutaneous T-cell Lymphomas: (Mycosis Fungoides, Sezary Syndrome): chemorefractory disease of > 2 prior regimens

Hodgkins Disease: refractory or persistent disease and not candidate for ASCT, or failed prior ASCT.

Peripheral T-cell Lymphoma

Exclusion Criteria:

* Age > 75 years and < 19 years
* progressive disease within 8 weeks of prior therapy or within 12 weeks after prior autologous stem cell transplantation
* Active CNS malignancy (patients with known positive CSF cytology or parenchymal lesions visible by CT or MRI)
* Fertile men or women unwilling to use appropriate contraceptive techniques during and for 12 months following treatment
* Females who are pregnant
* Patients who are HIV seropositive
* Active uncontrolled infection or immediate life-threatening condition at the time of enrollment
* Significant Organ dysfunction:

  1. Calculated Creatinine Clearance <55ml/min
  2. cardiac ejection fraction <40%, NYHA class II or greater cardiac disease.
  3. DLCO < 40% , FEV1/FVC ratio <50% predicted, or receiving supplementary continuous oxygen
  4. total bilirubin > 2x upper limit of normal (unless due to Gilberts disease or malignancy), ALT and AST 4x the upper limit of normal
* Karnofsky score <60%
* Patients with uncontrolled medical illnesses (e.g., uncontrolled systemic hypertension, diabetes)

Donor Inclusion Criteria:

* HLA genotypically matched relative
* siblings or first-degree relatives matched at HLA-A, B, or DR loci (6 antigen match) are acceptable donors
* HLA matched unrelated volunteer donor
* unrelated donor matched at HLA-A, B, or DR loci (6 antigen match) are acceptable donors
* One antigen mismatch related or unrelated donor will also be acceptable, molecular typing needs to be used at each H LA-A, B, or DR loci in case of mismatched unrelated donor.

Donor Exclusion Criteria:

* Identical twin
* Pregnancy
* HIV positive
* Serious Allergy to G-CSF
* Current serious systemic illness
* Failure to meet the UNMC or NMDP criteria for donors

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2000-12-08 (Actual); Primary Completion 2008-12-30 (Actual); Study Completion 2008-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Bociek, MD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Section of Oncology/Hematology, Omaha, Nebraska, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between November 2001 and February 2007 sixty eight patients were treated on this protocol and have been included in the analysis
Groups:
- Cohort I: Pentostatin to be administered intravenously on days -10, -9, and -8 at a dose of 4mg/m2/day
Period: Overall Study
Arm/Group | Cohort I
Started | 76
Completed | 68
Not Completed | 8
Not completed — Withdrawal by Subject | 2
Not completed — psychiatric instability | 1
Not completed — Adverse Event | 5

BASELINE CHARACTERISTICS:
Arm/Group | Cohort I
Number analyzed (Participants) | 76
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 71
  >=65 years | 5
Age, Continuous [Median (Full Range); unit: years] | 56 [21 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 47
Region of Enrollment [Number; unit: participants]
  United States | 76

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants With Chimerism: Full Donor Chimerism Defined as >95% Donor CD3+ Cell in Blood as Assessed by DNA Fingerprinting
Description: the efficacy of the regimen as determined by engraftment rate and establishment of donor hematopoietic chimerism at day +28 and day +70.
Time Frame: days +28 and +70
Measure: Median (Full Range); unit: percent of participants
Arm/Group | Cohort I
Number analyzed (Participants) | 68
percent of participants
  Day 28 | 85 [40 to 100]
  Day 70 | 90 [45 to 100]

2. Primary Outcome: Toxicity for the Combination of Pentostatin and Low Dose Total Body Irradiation (TBI)
Time Frame: Conditioning regimen to count recovery (D + 28 post transplant)
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort I
Number analyzed (Participants) | 68
Participants
  Absolute neutrophil count < 500/mm^3 | 40
  platelet count < 20,000/mm^3 | 29
  Grade 3 or 4 Fever | 2
  Grade 3 or 4 hypokalemia | 1
  Grade 3 or 4 bacteremia | 2
  Grade 3 or 4 infection | 6
  Grade 3 or 4 renal toxicity | 1
  Grade 3 or 4 thromboembolism | 1

3. Secondary Outcome: Incidence of Acute and Chronic Graft-versus-host Disease
Description: Incidence of acute and chronic graft-versus-host disease. Acute GVHD usually occurs during the first three months following transplant. Chronic GVHD usually develops after the third month post-transplant.
Time Frame: twice weekly until day 100 up to 1 year post transplant
Measure: Number; unit: Percent of Particpants
Arm/Group | Cohort I
Number analyzed (Participants) | 68
Percent of Particpants
  Acute GVHD | 31
  Chronic GVHD | 33

4. Secondary Outcome: Responses to Therapy
Description: event-free and overall survival at 12 months
Time Frame: every 6 mo. up to 2 years
Measure: Number; unit: Percent of Participants
Arm/Group | Cohort I
Number analyzed (Participants) | 68
Percent of Participants
  Event free survival | 52
  Overall survival | 59

5. Secondary Outcome: Kinetics of Immunologic Reconstitution
Description: Rate of return of immune cells after allogeneic transplantation
Time Frame: at day 100 post transplantation
Measure: Median (Full Range); unit: percentage of cells in peripheral blood
Groups:
- Study Baseline: T-cell count (CD3, CD4 and CD8 cells) prior to transplant
- Day + 28 Post Transplant: T-cell count (CD3, CD4 and CD8 cells) on Day + 28 post transplant. Measure of donor chimerism (donor CD3+ Cell in blood as assessed by DNA fingerprinting)
Arm/Group | Study Baseline | Day + 28 Post Transplant
Number analyzed (Participants) | 68 | 68
percentage of cells in peripheral blood
  CD3 cells | 13 [0.5 to 45] | 7 [0 to 28]
  CD4 cells | 5 [0.01 to 25] | 3.5 [0 to 13]
  CD8 cells | 5 [0 to 31] | 1.7 [0.02 to 8.3]

ADVERSE EVENTS:
Arm/Group | Cohort I
Serious Adverse Events (participants affected / at risk) | 26/76
Other Adverse Events (participants affected / at risk) | 0/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort I (N=76)
fever (General disorders) | 3 (3)
decreased WBC (Blood and lymphatic system disorders) | 9 (9)
decreased ANC (Blood and lymphatic system disorders) | 7 (7)
decreased hgb (Blood and lymphatic system disorders) | 1 (1)
decreased platelets (Blood and lymphatic system disorders) | 3 (3)
hypokalemia (Gastrointestinal disorders) | 1 (1)
decreased leukocyte (Blood and lymphatic system disorders) | 1 (1)
klebsiella (Cardiac disorders) | 1 (1)
reddened catheter site (Infections and infestations) | 1 (1)
herpes simplex (Immune system disorders) | 1 (1)
Yeast infection (Renal and urinary disorders) | 1 (1)
increased LDH (Hepatobiliary disorders) | 1 (1)
pulmonary embolism (Blood and lymphatic system disorders) | 1 (1)
azotemia (Renal and urinary disorders) | 1 (1)
atubular necrosis (Renal and urinary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No